CLINICAL TRIAL: NCT07229716
Title: Study on the Drug Interactions of HRS-9813, Pirfenidone and Nintedanib in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-9813-105
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-9813 Capsule or Nintedanib Soft Capsules or Pirfenidone Tablets Group (Experimental)
  Interventions: Drug: HRS-9813 Capsule; Drug: Nintedanib Soft Capsules; Drug: Pirfenidone Tablets

INTERVENTIONS:
Drug: HRS-9813 Capsule — HRS-9813 capsule, specified dose on specified days.
Drug: Nintedanib Soft Capsules — Nintedanib soft capsules, specified dose on specified days.
Drug: Pirfenidone Tablets — Pirfenidone tablets, specified dose on specified days.

SUMMARY:
This study aims to evaluate the interaction of oral HRS-9813 capsules with pirfenidone and nintedanib on the pharmacokinetics of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of the related activities of this trial, and be able to understand the procedures and methods of this trial. Also, be willing to strictly follow the clinical trial protocol to complete this trial.
2. Aged 18-45 years.
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 19 - 28 kg/m2 (including both endpoints).
4. Sign the informed consent form and, within 28 days after the last administration of the trial drug, have no intention of having children and agree to adopt non-drug methods of effective contraception, and have no plans for sperm donation or egg donation.

Exclusion Criteria:

1. Those who are allergic to the study drugs (HRS-9813 capsules, nintedanib or pirfenidone), or any components of the study drugs, or have an allergic constitution (such as individuals with asthma, allergic rhinitis, or eczema).
2. Those subjects who, in the judgment of the researchers, have any conditions or diseases that may affect the absorption, metabolism, and/or excretion of the study drug.
3. Those who participated in any clinical trial of other drugs or medical devices within the previous 3 months before the screening period or baseline period, or those whose exposure to the drug is still within 5 half-lives during the study period (whichever is longer).
4. During the screening period or baseline period, the sitting systolic blood pressure was less than 90 mmHg or the sitting diastolic blood pressure was less than 60 mmHg.
5. During the screening period, any one of the following being positive: hepatitis B surface antigen (HBsAg), human immunodeficiency virus antibody, Treponema pallidum antibody or hepatitis C virus antibody.
6. Pregnant or lactating women, or those whose blood pregnancy test results in the screening or baseline phase are positive.
7. Those who have a history of blood donation within 8 weeks before the screening period or the baseline period, or have suffered from severe blood loss (blood loss ≥ 400 mL), or have received blood transfusion within 4 weeks before the screening period or the baseline period; or those who plan to donate blood during the trial.
8. Those who were vaccinated within the two weeks prior to the screening period or the baseline period, or those who plan to receive the vaccine during the trial process.
9. Those who have special dietary requirements and cannot follow the uniform diet.
10. Those who have difficulty swallowing, have problems with venous blood collection, or whose physical condition does not allow for intensive blood sampling.
11. Those who have had severe infections, severe trauma or undergone heavy manual surgery within 3 months before the screening period or baseline period; Or those who plan to undergo surgery during the trial period.
12. During the screening period or baseline period, for those with abnormal 12-lead electrocardiogram results and clinical significance, the QTcB of men was > 450ms and that of women was > 460 ms.
13. Those who have a history of smoking (smoking more than 5 cigarettes per day on average) within 3 months before the screening period or baseline period, or those who have a smoking history within 4 weeks before the screening period or baseline period, or those who cannot stop using any tobacco products during the trial period.
14. Those who have a history of drug use or drug abuse/dependence before the screening period or baseline period; Or those with positive urine test results during the baseline period.
15. Those who consumed excessive amounts of tea, coffee or caffeinated beverages (an average of more than 8 cups per day, 250 mL per cup) within 6 months prior to the screening period or baseline period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | From Day 1 to Day 24.
Area under the concentration curve from time 0 to extrapolated infinite time (AUC0-inf) | From Day 1 to Day 24.
Area under the concentration curve from time 0 to time of last quantifiable concentration (AUC0-tau) | From Day 1 to Day 24.
Area under the concentration curve from time 0 to time t (AUC0-t) | From Day 1 to Day 24.

SECONDARY OUTCOMES:
Accumulative excretion rate (Ae) | Day 1, Day 19 and Day 20.
Fractional excretion (Fe) | Day 1, Day 19 and Day 20.
Renal clearance (CLr) | Day 1, Day 19 and Day 20.
Adverse events (AEs) | From Day 1 to Day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Fourth Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided